CLINICAL TRIAL: NCT02176148
Title: Cutaneous Lupus Medication Experience Study
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00026573
Record Dates: First submitted 2014-06-24; First posted 2014-06-26 (Estimated); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Cutaneous Lupus
Keywords: cutaneous lupus; systemic lupus; systemic therapy; medication
MeSH Terms: interventions — Fluocinonide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lupus control standard-of-care: Each person enrolled will be given fluocinonide 0.05% cream to apply twice daily to active areas.
  Interventions: Drug: fluocinonide 0.05% cream

INTERVENTIONS:
Drug: fluocinonide 0.05% cream

SUMMARY:
Cutaneous lupus is a chronic, relapsing, auto-immune skin disease that can have many presentations. Its effect on physical appearance greatly affects patients' quality of life. In addition, 10% of patients with cutaneous lupus will develop systemic lupus. Topical therapies are the mainstay of cutaneous lupus treatment; however patients often find these treatments to be messy, inconvenient, or ineffective. In addition, for more severe disease patients are often placed on concurrent systemic therapies. The primary hypothesis of our study is that poor adherence contributes to poor treatment outcomes in patients with cutaneous lupus.

DETAILED DESCRIPTION:
Cutaneous lupus is a chronic, relapsing auto-immune disease that negatively impacts patients' quality of life. As there are many safe topical therapies that require daily use to be effective, and adherence to medication remains a common problem in dermatology, it is worthwhile to reliably measure adherence to medication in patients with cutaneous lupus. By elucidating barriers to effective control of cutaneous lupus with topical medications, we can improve patient care and guide interventions that will avoid the use of systemic therapy which often has more side effects.

The primary aim is to determine adherence to topical and systemic lupus treatment. Subjects will receive standard of care therapy (low potency and high potency topical corticosteroids) and systemic therapy when clinically appropriate. Adherence to medications will be monitored electronically in all subjects. The following hypothesis is to be tested: Non-adherence to topical and systemic medication contributes to treatment failure in patients with cutaneous lupus.

ELIGIBILITY:
Inclusion Criteria:

* Any male or female 12 years or older of age with a diagnosis of cutaneous lupus by a dermatologist
* Capable of understanding and willing to provide a signed and dated written voluntary informed consent before any protocol specific procedures are performed
* Able to complete the study and comply with study instructions, including attending all study visits

Exclusion Criteria:

* Individuals younger than 12 years of age
* Known allergy or sensitivity to study medication
* Inability to complete all study-related visits
* Introduction of any other prescription medication, topical or systemic, for cutaneous lupus while participating in the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Dermatology clinic patients with a diagnosis of active cutaneous lupus confirmed by a dermatologist
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2014-12; Primary Completion 2020-12-04 (Actual); Study Completion 2020-12-04 (Actual)

PRIMARY OUTCOMES:
Change in Adherence Measures | up to 6 month
  There will be interim measures taken after the baseline measure at month 1, month 3, and at end point month 6.

SECONDARY OUTCOMES:
Disease Severity Measures | 6 months
  Assessments will be taken at baseline, month 1, month 3, and at end point month 6.
  1. Change in cutaneous lupus severity, measured by the Investigator's Global Assessment of severity (IGA) and Cutaneous Lupus Erythematosus Disease Area Severity Index (CLASI) scales.
  2. Factors that affect adherence to lupus treatment, including physician trust, trust in the medication, and confidence in the treatment plan which will be measured with the Wake Forest University Physician Trust Scale (WFUPTS). and the Treatment Satisfaction Questionnaire for Medication (TSQM).

CONTACTS AND LOCATIONS:
Overall Officials: William W Huang, MD, MPH, FAAD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University School of Medicine - Department of Dermatology, Winston-Salem, North Carolina, United States